CLINICAL TRIAL: NCT07121088
Title: Comparative Effectiveness Study of Traditional Chinese Medicine Intervention in Ischemic Cerebrovascular Disease Comorbid With Diabetes Mellitus
Brief Title: Traditional Chinese Medicine Intervention for Ischemic Cerebrovascular Disease and Diabetes Mellitus: An Efficacy Comparative Study
Acronym: TIDES
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023ZD0505604
Record Dates: First submitted 2025-07-04; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Cerebral Infarction; Diabetes Mellitus
Keywords: diabetes mellitus; ischemic cerebral infarction; Chuanzhitongluo capsule
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chuanzhitongluo capsule+Standard Treatment (Experimental): On the basis of standard treatment, a combined treatment plan of TCM universal treatment and syndrome-specific treatment was given.
  TCM universal treatment plan:
  (Intensive treatment) Chuanzhi Tongluo Capsules (Lunan Pharmaceutical), 4 capsules each time, orally, 3 times a day; administration from day 1 to day 14 of the disease.
  (Sequential treatment) Chuanzhi Tongluo Capsules (Lunan Pharmaceutical), 2 capsules each time, orally, 3 times a day; administration from day 15 to day 365.
  TCM decoction: Individualized herbal decoction based on TCM diagnosis (four diagnostic methods), administered for 14 days during intensive phase.
  Interventions: Drug: (Intensive treatment) Chuanzhi Tongluo Capsules; Drug: (Sequential treatment) Chuanzhi Tongluo Capsules; Drug: TCM Syndrome Differentiation Decoction
- Standard Treatment Only (Active Comparator): Guideline-based treatment for cerebral infarction with diabetes: aspirin (100 mg/day) + clopidogrel (75 mg/day) + atorvastatin (20 mg/day) + metformin (500 mg bid). Other antiplatelet/antidiabetic drugs may be added per clinician discretion.
  Interventions: Other: Standard Treatment (Guideline-Based)

INTERVENTIONS:
Drug: (Intensive treatment) Chuanzhi Tongluo Capsules — 4 capsules each time, orally, 3 times a day; administration from day 1 to day 14 of the disease.
  Arms: Chuanzhitongluo capsule+Standard Treatment
Other: Standard Treatment (Guideline-Based) — Combination therapy including: 1. Antiplatelet: aspirin 100 mg/day + clopidogrel 75 mg/day. 2. Lipid-lowering: atorvastatin 20 mg/day. 3. Antidiabetic: metformin 500 mg bid (max 2000 mg/day). *Doses may be adjusted per local guidelines or patient tolerance.
  Arms: Standard Treatment Only
Drug: (Sequential treatment) Chuanzhi Tongluo Capsules — 2 capsules each time, orally, 3 times a day; administration from day 15 to day 365.
  Arms: Chuanzhitongluo capsule+Standard Treatment
Drug: TCM Syndrome Differentiation Decoction — Individualized herbal decoction based on TCM diagnosis (four diagnostic methods), administered for 14 days during intensive phase.
  Arms: Chuanzhitongluo capsule+Standard Treatment

SUMMARY:
The objective of this observational study is to understand the long-term effects of traditional Chinese medicine (TCM) intervention on patients with cerebral infarction onset within <48 hours and comorbid diabetes. The primary question it aims to address is:

Can long-term TCM intervention for the treatment of ischemic cerebrovascular disease comorbid with diabetes improve patients' neurological deficits and self-care ability? Participants receiving TCM intervention (universal treatment combined with syndrome-specific treatment) as part of routine cerebrovascular disease management will undergo follow-up assessments at 30 days, 90 days, 6 months, and 12 months within 1 year to evaluate neurological status (e.g., mRS score, NIHSS score) and quality of life indicators.

DETAILED DESCRIPTION:
The population with ischemic cerebrovascular disease (ICVD) comorbid with diabetes is growing, characterized by high mortality, disability, and recurrence rates of vascular events, with a lack of effective treatments. There are 529 million diabetic patients worldwide and 129 million in China, among which 43 million have comorbid vascular diseases; China has approximately 10 million ischemic stroke patients, with 4.5 million comorbid diabetes. Diabetes increases the risk of ischemic stroke, and the proportion of deaths related to diabetic cerebrovascular diseases has risen significantly. Polypharmacy also raises the risk of adverse drug interactions, imposing a heavy medical burden.

The pathological mechanism aligns with the TCM theory of "toxin damaging collaterals": Diabetes-induced glucose/lipid metabolism disorders and activation of the renin-angiotensin-aldosterone system cause systemic vascular endothelial dysfunction and atherosclerosis. Macrovascular lesions mainly involve atherosclerosis, while microvascular lesions include endothelial damage and microcirculatory disorders, with core mechanisms involving energy metabolism abnormalities and mitochondrial dysfunction. TCM holds that "excessive pathogens transform into toxins," and toxin-induced collateral damage disrupts structure and function, consistent with the above pathology. Thus, "detoxification and collaterals dredging" (combining qi-nourishing, blood-activating, and stasis-removing) is the core therapeutic principle.

Chuanzhi Tongluo Capsules (Lunan Pharmaceutical), a Shandong famous brand with annual sales over 100 million yuan, exert effects of promoting blood circulation and dredging collaterals, reducing inflammation and improving microcirculation. This project explores a TCM program combining "acute-phase intensive treatment + recovery-phase sequential treatment" and "universal + syndrome-specific treatment." Entitled Comparative Efficacy Study of TCM Intervention in ICVD Comorbid with Diabetes, this Phase IV trial spans 4 years, adopting a multi-center real-world non-randomized controlled design. It will enroll 3,666 patients with acute cerebral infarction (onset <48h) comorbid diabetes across 50 centers. The control group receives standard secondary prevention of cerebrovascular disease and hypoglycemic treatment; the trial group adds Chuanzhi Tongluo Capsules (4 capsules thrice daily for 14 days, then 2 capsules thrice daily for 1 year) plus syndrome-specific treatment (5 TCM syndromes with corresponding herbs for 14 days).

Inclusion criteria: ≥18 years old, meeting diabetes/acute ischemic stroke criteria, and TCM "toxin damaging brain collaterals" syndrome. Exclusions: hemorrhagic transformation, large infarction, type 1 diabetes, etc. The primary endpoint is the proportion of patients with mRS 0-2 at 90 days. Secondary endpoints include 1-year BARC type III/V major bleeding, MACCE, all-cause mortality, diabetic microvascular lesions (renal indices), mRS, MMSE, and EQ-5D-5L at 6/12 months. Data are managed via EpiData and analyzed with SAS, using chi-square test, t-test, and rank sum test, with 90% statistical power (α=0.05, β=0.10). The trial aims to establish a "disease-syndrome combined" long-term intervention model, expanding TCM applicability and evidence generalization.

English Abbreviation The population with ischemic cerebrovascular disease (ICVD) comorbid with diabetes is growing, with high mortality, disability, and recurrence rates of vascular events, and a lack of effective treatments. Globally, there are 529 million diabetic patients, including 129 million in China, among whom 43 million have comorbid vascular diseases; China has ~10 million ischemic stroke patients, with ~4.5 million comorbid diabetes. Diabetes elevates ischemic stroke risk, and related deaths are increasing, while polypharmacy raises adverse interactions and medical burdens.

Pathologically, it aligns with TCM's "toxin damaging collaterals" theory: Diabetes-induced metabolic disorders and systemic vascular activation cause endothelial dysfunction and atherosclerosis (macrovascular lesions) and microcirculatory disorders (microvascular lesions), involving energy metabolism and mitochondrial dysfunction. TCM holds toxins damage collaterals, disrupting structure/function, consistent with the pathology, so "detoxification and collaterals dredging" (combining qi-nourishing, blood-activating) is key.

Chuanzhi Tongluo Capsules (Lunan Pharmaceutical), a Shandong famous brand with annual sales over ¥100 million, improve circulation and reduce inflammation. This Phase IV trial (4 years) uses a multi-center real-world non-randomized design, enrolling 3,666 patients (onset <48h) across 50 centers. The control group receives standard care; the trial group adds Chuanzhi Tongluo Capsules (intensive: 4 caps thrice daily for 14 days; sequential: 2 caps thrice daily for 1 year) plus syndrome-specific herbs for 5 TCM syndromes.

Inclusion: ≥18 years, meeting diabetes/ischemic stroke criteria, and "toxin damaging brain collaterals" syndrome. Exclusions: hemorrhagic transformation, large infarction, type 1 diabetes, etc. Primary endpoint: 90-day mRS 0-2 proportion. Secondary endpoints: 1-year BARC III/V bleeding, MACCE, mortality, diabetic microvascular lesions, mRS, MMSE, EQ-5D-5L at 6/12 months. Analyzed via EpiData and SAS (chi-square, t-test, rank sum test) with 90% power (α=0.05, β=0.10). It aims to establish a "disease-syndrome combined" model, expanding TCM applicability and evidence generalization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, regardless of gender.
2. Previously diagnosed with diabetes, or with an unknown medical history, meeting the WHO 2023 diagnostic criteria for type 2 diabetes, including any of the following:

   * Fasting blood glucose ≥ 7.0 mmol/L.
   * 2-hour postprandial blood glucose ≥ 11.1 mmol/L.
   * Glycated hemoglobin ≥ 6.5%.
3. Acute cerebral infarction meets the diagnostic criteria of *Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2023*:

   * Acute onset.
   * Focal neurological deficits, with a few cases showing global neurological deficits.
   * The presence of a responsible lesion on imaging or symptoms/signs persisting for more than 24 hours.
   * Exclusion of non-vascular etiologies.
   * Exclusion of intracerebral hemorrhage by brain CT/MRI.
4. Onset of cerebral infarction < 48 hours.
5. TCM syndrome conforms to the "toxin damaging brain collaterals" syndrome (referring to the diagnostic criteria (draft) of *Research on the Diagnostic Criteria for the Syndrome of Mutual Binding of Stasis and Toxin in Ischemic Cardiovascular and Cerebrovascular Diseases* (Ju Jianqing et al., 2023)).
6. Modified Rankin Scale (mRS) before onset: 0 - 1 point.
7. National Institutes of Health Stroke Scale (NIHSS) at admission: 4 - 24 points.
8. Signed informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3666 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome indicator | 90days
  The proportion of patients with mRS score 0-2 at 90 days

SECONDARY OUTCOMES:
BARC Type III and V Major Bleeding (Incidence %) | 1year
  The percentage of patients meeting the following criteria: Type IIIa is overt bleeding with a hemoglobin drop of 3-<5 g/dL or requiring transfusion; Type IIIb is a hemoglobin drop of >5 g/dL, cardiac tamponade, bleeding requiring surgical intervention (excluding dental/nasal/skin/hemorrhoidal bleeding), or requiring intravenous vasoactive drugs; Type IIIc is intracranial/spinal hemorrhage (excluding microhemorrhage/hemorrhagic transformation); Type V is fatal bleeding.
1-Year Major Adverse Cardiovascular and Cerebrovascular Events (MACCEs) (Cumulative Incidence %) | 1year
  The percentage of patients who experience major adverse cardiovascular and cerebrovascular events (in accordance with international criteria: including myocardial infarction, recurrent stroke, cardiovascular death, etc.) within 1 year.
1-Year All-Cause Mortality (Mortality Rate %) | 1year
  The percentage of patients who die from any cause within 1 year after treatment.

OTHER OUTCOMES:
Rate of Change in eGFR (mL/min/1.73 m²/year) | Baseline, 6 months, 12 months
  Estimated glomerular filtration rate (eGFR) calculated using CKD-EPI formula. Annualized rate of change derived from serial measurements at baseline, 6, and 12 months.
12-month Renal Composite Endpoint | 12 months
  Composite of: 1) Sustained ≥50% decline in eGFR from baseline; 2) Sustained eGFR <15 mL/min/1.73 m²; 3) Initiation of long-term dialysis or renal transplantation.
Rate of Change in UACR (mg/g/year) | Baseline, 6 months, 12 months
  Urine albumin-to-creatinine ratio (UACR) measured from first-morning void samples. Annualized rate of change calculated from baseline, 6, and 12-month data.
Change in Tubular Markers (α1-MG, β2-MG, NAG) at 12 Months | Baseline, 12 months
  Urinary biomarkers of tubular injury: α1-microglobulin (α1-MG), β2-microglobulin (β2-MG), and N-acetyl-β-D-glucosaminidase (NAG). Concentrations measured by immunoturbidimetry (α1-MG, β2-MG) and enzymatic assay (NAG).

IPD SHARING:
Plan to Share IPD: Undecided